CLINICAL TRIAL: NCT02053831
Title: GalaFlex Mesh in Facelift
Status: Completed | Type: Observational
Sponsor: C. R. Bard (Industry)
Collaborators: Tepha, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-1040
Record Dates: First submitted 2014-01-31; First posted 2014-02-04 (Estimated); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Superficial Musculoaponeurotic System (SMAS) Procedure
Keywords: plastic surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In this post market study a resorbable mesh (GalaFLEX) will be used to reinforce the lifted and imbricated SMAS along the suture lines and spread the load of the SMAS along a greater surface area. GalaFLEX mesh is comprised of resorbable 4-hydroxybutyrate fibers.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to understand the risks and benefits of participating in the study and must be willing to sign and date the Informed Consent Form for this study approved by the Institutional Review Board (IRB.)
* Be at least 21 years of age.
* Be willing and able to comply with the requirements of the protocol.
* Be willing to refrain from participating in any other investigational interventional study while enrolled in this study.
* Female subjects must have a negative pregnancy test within the last 24 hours timeline and have no intentions of becoming pregnant during participation in the study, or be sterilized.

Exclusion Criteria:

* Subject is unwilling or unable to give written consent to participate in the investigation or unable to comply with the requirements of the protocol.
* Subject has known severe allergies manifested by a history of anaphylaxis, or history or presence of severe multiple allergies.
* Subject has any serious skin disease, e.g., Eczema and psoriasis of the face, severe rosacea, scleroderma, local infections and severe acne.
* Subjects has diabetes, coagulation disorders, connective tissue disorders, lipodystrophy, or other serious systemic disease.
* Active herpes labialis
* Subject is infected with HIV and/or received or may receive immunosuppressive therapy over the course of the study (such as rheumatoid arthritis).
* Received any experimental drug or device within the previous three months.
* Known alcohol or drug abuser.
* Female subject who is pregnant or lactating or intending to become pregnant during the period of the study, or who would not use an adequate method of contraception (contraceptive pill, intra-uterine device) for the duration of the study.
* Possesses any psychological condition, or is under treatment for any condition which, in the opinion of the Investigator and/or consulting physicians(s),would constitute an unwarranted risk.
* Presents with severe jowling or severe cervical skin redundancy.
* Subject is currently a smoker or is a prior smoker who quit in the last 12 months.
* Active abscess or infection
* Currently involved with claims for, or is accepting, workers compensation
* Currently engaged in medical malpractice litigation.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinics
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2011-11; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Physician Satisfaction | 1 year
  Investigator satisfaction will be judged by ease of product use, successful reinforcement, and total time for procedure to be completed.

SECONDARY OUTCOMES:
Patient Satisfaction | 1 year
  Patient satisfaction will be judged by the difference between pre- and post-surgery answers to Quality of Life questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Arikha Moses, Ph.D, Study Director — Chief Scientific Officer, Founder
Locations (3):
- United States (3):
  - Ponte Vedra Plastic Surgery, Ponte Vedra Beach, Florida
  - The Few Institute for Aesthetic Plastic Surgery, Chicago, Illinois
  - Eye and Ear Institute, Chicago, Illinois